CLINICAL TRIAL: NCT02906332
Title: A Phase II Trial of the Anti -PD-1 Monoclonal Antibody Pembrolizumab (MK-3475) + Lenalidomide + Dexamethasone as Post Autologous Transplant Consolidation in Patients With High-risk Multiple Myeloma
Brief Title: Pembrolizumab + Lenalidomide Post Autologous Stem Cell Transplant (ASCT) in High-risk Multiple Myeloma (MM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA Hold Due to Updated Risks
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2016-0262
Record Dates: First submitted 2016-05-26; First posted 2016-09-20 (Estimated); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — pembrolizumab; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab + lenalidomide (Experimental): This is an open label study.
  * Pembrolizumab 200 mg IV every 3 weeks and lenalidomide 25 mg po daily x 14 days and dexamethasone 40 mg po once weekly for a 21-day cycle x 2 cycles.
  * This is followed by pembrolizumab 200 mg every 3 weeks and lenalidomide 25 mg po daily x 14 days for a 21-day cycle x 2 cycles for a total of 4 cycles.
  Interventions: Drug: Pembrolizumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV every 3 weeks x 2 cycles. This is followed by followed by pembrolizumab 200 mg IV every 3 weeks for 2 additional cycles.
  Other Names: Keytruda
Drug: Lenalidomide — Lenalidomide 25 mg po daily x 14 days once weekly for a 21-day cycle x 2 cycles. This is followed by lenalidomide 25 mg po daily x 14 days for a 21-day cycle x 2 cycles for 2 additional cycles.
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone 40 mg po once weekly for a 21-day cycle x 2 cycles only.
  Other Names: Decadron

SUMMARY:
This is an open-label, Phase II, single center trial of pembrolizumab (MK-3475), lenalidomide and dexamethasone in subjects with high risk Multiple Myeloma (hrMM) post high-dose chemotherapy with autologous stem cell transplantation (ASCT).

Patients with high-risk MM defined as those with one of the following abnormalities who have undergone induction therapy followed by single or tandem melphalan -based ASCT will be considered eligible.

DETAILED DESCRIPTION:
The primary objectives of this trial are to establish the progression free survival (PFS) of ASCT followed by consolidative therapy with pembrolizumab plus lenalidomide and dexamethasone and to evaluate the safety of pembrolizumab plus lenalidomide and dexamethasone following ASCT. The immunological analysis of cells and cytokines pre and post-therapy will be determined from patient bone marrow aspirate and peripheral blood samples as exploratory objectives. The overall composition of the gut microbiome will also be determined in patient stool samples.

Patients will be followed by response, EFS/PFS/OS and safety endpoints on an every 3 week basis. Bone marrow aspirate specimens will be obtained at screening and at completing of the study and peripheral blood specimens will be obtained on a monthly basis to evaluate in correlative studies.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age on day of signing informed consent.
* Has a confirmed diagnosis of MM based on standard criteria. (See Appendix 2 for MM Diagnostic Criteria.)
* Is between 60 and 180 days from peripheral blood autologous stem cell transplant.
* At diagnosis, had MM with measurable disease, defined as:
* A monoclonal immunoglobulin spike on serum electrophoresis of at least 0.5 g/dL and/or
* Urine monoclonal levels of at least 200 mg/24 hours
* For subjects without measurable serum and urine M-protein levels, an abnormal free light chain (FLC) ratio (normal value 0.26 - 1.65) with involved FLC ≥10 mg/dL
* Radiographic evidence of disease for those without measurable M-spike or free light chains.
* Has high-risk MM, which must be present at the time of diagnosis, and defined by:

  * International Staging System (ISS) stage 3 (See Appendix 3 for ISS Staging), and/or
  * Deletion 13q by cytogenetics, and/or
  * 1q amplification, 1p deletion, p53 deletions (17p deletions), t(4;14), t(14;16), t(14;20), hypodiploidy, and/or
  * High-risk gene expression profile (GEP) scores
* Be able to provide a newly obtained bone marrow aspirate/biopsy material for biomarker analysis and disease assessment.
* Have a performance status of ≤2 on the ECOG Performance Scale (See Appendix 4).
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 28 days of treatment initiation.
* All subjects must agree to follow the regional requirements for lenalidomide counseling, pregnancy testing, and birth control; and be willing and able to comply with the regional requirements (for example, periodic pregnancy tests, safety labs, etc.).
* Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 10-14 days prior to and again within 24 hours prior to receiving the first dose of pembrolizumab (MK-3475), lenalidomide and dexamethasone or pembrolizumab (MK-3475) and lenalidomide. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female subjects of childbearing potential should agree to ongoing pregnancy testing.
* Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 4.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 2 years.
* Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential even if they have had a successful vasectomy starting with the first dose of study therapy through 120 days after the last dose of study therapy.
* Subject is able to swallow capsules and is able to take or tolerate oral medications on a continuous basis.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be used at the investigator's discretion.
* Has received an allogeneic stem cell transplant.
* Has received any myeloma-directed therapy after ASCT.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Progressive disease from autologous transplantation at the time of screening
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring intravenous systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noa Biran, M.D., Principal Investigator — Hackensack Meridian Health
Locations (1):
- John Theurer Cancer Center-Hackensack Meridian Health, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taur Y, Jenq RR, Ubeda C, van den Brink M, Pamer EG. Role of intestinal microbiota in transplantation outcomes. Best Pract Res Clin Haematol. 2015 Jun-Sep;28(2-3):155-61. doi: 10.1016/j.beha.2015.10.013. Epub 2015 Oct 22. PMID 26590773
- [Background] Viaud S, Saccheri F, Mignot G, Yamazaki T, Daillere R, Hannani D, Enot DP, Pfirschke C, Engblom C, Pittet MJ, Schlitzer A, Ginhoux F, Apetoh L, Chachaty E, Woerther PL, Eberl G, Berard M, Ecobichon C, Clermont D, Bizet C, Gaboriau-Routhiau V, Cerf-Bensussan N, Opolon P, Yessaad N, Vivier E, Ryffel B, Elson CO, Dore J, Kroemer G, Lepage P, Boneca IG, Ghiringhelli F, Zitvogel L. The intestinal microbiota modulates the anticancer immune effects of cyclophosphamide. Science. 2013 Nov 22;342(6161):971-6. doi: 10.1126/science.1240537. PMID 24264990
- [Background] Iida N, Dzutsev A, Stewart CA, Smith L, Bouladoux N, Weingarten RA, Molina DA, Salcedo R, Back T, Cramer S, Dai RM, Kiu H, Cardone M, Naik S, Patri AK, Wang E, Marincola FM, Frank KM, Belkaid Y, Trinchieri G, Goldszmid RS. Commensal bacteria control cancer response to therapy by modulating the tumor microenvironment. Science. 2013 Nov 22;342(6161):967-70. doi: 10.1126/science.1240527. PMID 24264989
- [Background] Vetizou M, Pitt JM, Daillere R, Lepage P, Waldschmitt N, Flament C, Rusakiewicz S, Routy B, Roberti MP, Duong CP, Poirier-Colame V, Roux A, Becharef S, Formenti S, Golden E, Cording S, Eberl G, Schlitzer A, Ginhoux F, Mani S, Yamazaki T, Jacquelot N, Enot DP, Berard M, Nigou J, Opolon P, Eggermont A, Woerther PL, Chachaty E, Chaput N, Robert C, Mateus C, Kroemer G, Raoult D, Boneca IG, Carbonnel F, Chamaillard M, Zitvogel L. Anticancer immunotherapy by CTLA-4 blockade relies on the gut microbiota. Science. 2015 Nov 27;350(6264):1079-84. doi: 10.1126/science.aad1329. Epub 2015 Nov 5. PMID 26541610
- [Background] Sivan A, Corrales L, Hubert N, Williams JB, Aquino-Michaels K, Earley ZM, Benyamin FW, Lei YM, Jabri B, Alegre ML, Chang EB, Gajewski TF. Commensal Bifidobacterium promotes antitumor immunity and facilitates anti-PD-L1 efficacy. Science. 2015 Nov 27;350(6264):1084-9. doi: 10.1126/science.aac4255. Epub 2015 Nov 5. PMID 26541606
- [Background] Disis ML. Immune regulation of cancer. J Clin Oncol. 2010 Oct 10;28(29):4531-8. doi: 10.1200/JCO.2009.27.2146. Epub 2010 Jun 1. PMID 20516428
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Sharpe AH, Freeman GJ. The B7-CD28 superfamily. Nat Rev Immunol. 2002 Feb;2(2):116-26. doi: 10.1038/nri727. PMID 11910893
- [Background] Brown JA, Dorfman DM, Ma FR, Sullivan EL, Munoz O, Wood CR, Greenfield EA, Freeman GJ. Blockade of programmed death-1 ligands on dendritic cells enhances T cell activation and cytokine production. J Immunol. 2003 Feb 1;170(3):1257-66. doi: 10.4049/jimmunol.170.3.1257. PMID 12538684
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Thompson RH, Dong H, Lohse CM, Leibovich BC, Blute ML, Cheville JC, Kwon ED. PD-1 is expressed by tumor-infiltrating immune cells and is associated with poor outcome for patients with renal cell carcinoma. Clin Cancer Res. 2007 Mar 15;13(6):1757-61. doi: 10.1158/1078-0432.CCR-06-2599. PMID 17363529
- [Background] Talmadge JE, Donkor M, Scholar E. Inflammatory cell infiltration of tumors: Jekyll or Hyde. Cancer Metastasis Rev. 2007 Dec;26(3-4):373-400. doi: 10.1007/s10555-007-9072-0. PMID 17717638
- [Background] Usubutun A, Ayhan A, Uygur MC, Ozen H, Toklu C, Ruacan S. Prognostic factors in renal cell carcinoma. J Exp Clin Cancer Res. 1998 Mar;17(1):77-81. PMID 9646237
- [Background] Al-Shibli KI, Donnem T, Al-Saad S, Persson M, Bremnes RM, Busund LT. Prognostic effect of epithelial and stromal lymphocyte infiltration in non-small cell lung cancer. Clin Cancer Res. 2008 Aug 15;14(16):5220-7. doi: 10.1158/1078-0432.CCR-08-0133. PMID 18698040
- [Background] Deschoolmeester V, Baay M, Van Marck E, Weyler J, Vermeulen P, Lardon F, Vermorken JB. Tumor infiltrating lymphocytes: an intriguing player in the survival of colorectal cancer patients. BMC Immunol. 2010 Apr 12;11:19. doi: 10.1186/1471-2172-11-19. PMID 20385003
- [Background] Diez M, Pollan M, Enriquez JM, Dominguez P, Santana A, Tobaruela E, Muguerza JM, Arrieta F, Rodriguez A, Ruiz A. Histopathologic prognostic score in colorectal adenocarcinomas. Anticancer Res. 1998 Jan-Feb;18(1B):689-94. PMID 9584053
- [Background] Galon J, Costes A, Sanchez-Cabo F, Kirilovsky A, Mlecnik B, Lagorce-Pages C, Tosolini M, Camus M, Berger A, Wind P, Zinzindohoue F, Bruneval P, Cugnenc PH, Trajanoski Z, Fridman WH, Pages F. Type, density, and location of immune cells within human colorectal tumors predict clinical outcome. Science. 2006 Sep 29;313(5795):1960-4. doi: 10.1126/science.1129139. PMID 17008531
- [Background] Hiraoka N. Tumor-infiltrating lymphocytes and hepatocellular carcinoma: molecular biology. Int J Clin Oncol. 2010 Dec;15(6):544-51. doi: 10.1007/s10147-010-0130-1. Epub 2010 Oct 6. PMID 20924634
- [Background] Nobili C, Degrate L, Caprotti R, Franciosi C, Leone BE, Trezzi R, Romano F, Uggeri F, Uggeri F. Prolonged survival of a patient affected by pancreatic adenocarcinoma with massive lymphocyte and dendritic cell infiltration after interleukin-2 immunotherapy. Report of a case. Tumori. 2008 May-Jun;94(3):426-30. doi: 10.1177/030089160809400323. PMID 18705415
- [Background] Hodi FS, Dranoff G. The biologic importance of tumor-infiltrating lymphocytes. J Cutan Pathol. 2010 Apr;37 Suppl 1(0 1):48-53. doi: 10.1111/j.1600-0560.2010.01506.x. PMID 20482675
- [Background] Kloor M. Lymphocyte infiltration and prognosis in colorectal cancer. Lancet Oncol. 2009 Sep;10(9):840-1. doi: 10.1016/S1470-2045(09)70245-1. No abstract available. PMID 19717085
- [Background] Hillen F, Baeten CI, van de Winkel A, Creytens D, van der Schaft DW, Winnepenninckx V, Griffioen AW. Leukocyte infiltration and tumor cell plasticity are parameters of aggressiveness in primary cutaneous melanoma. Cancer Immunol Immunother. 2008 Jan;57(1):97-106. doi: 10.1007/s00262-007-0353-9. Epub 2007 Jun 30. PMID 17602225
- [Background] Lee HE, Chae SW, Lee YJ, Kim MA, Lee HS, Lee BL, Kim WH. Prognostic implications of type and density of tumour-infiltrating lymphocytes in gastric cancer. Br J Cancer. 2008 Nov 18;99(10):1704-11. doi: 10.1038/sj.bjc.6604738. Epub 2008 Oct 21. PMID 18941457
- [Background] Leffers N, Gooden MJ, de Jong RA, Hoogeboom BN, ten Hoor KA, Hollema H, Boezen HM, van der Zee AG, Daemen T, Nijman HW. Prognostic significance of tumor-infiltrating T-lymphocytes in primary and metastatic lesions of advanced stage ovarian cancer. Cancer Immunol Immunother. 2009 Mar;58(3):449-59. doi: 10.1007/s00262-008-0583-5. Epub 2008 Sep 13. PMID 18791714
- [Background] Nishimura H, Honjo T, Minato N. Facilitation of beta selection and modification of positive selection in the thymus of PD-1-deficient mice. J Exp Med. 2000 Mar 6;191(5):891-8. doi: 10.1084/jem.191.5.891. PMID 10704469
- [Background] Liotta F, Gacci M, Frosali F, Querci V, Vittori G, Lapini A, Santarlasci V, Serni S, Cosmi L, Maggi L, Angeli R, Mazzinghi B, Romagnani P, Maggi E, Carini M, Romagnani S, Annunziato F. Frequency of regulatory T cells in peripheral blood and in tumour-infiltrating lymphocytes correlates with poor prognosis in renal cell carcinoma. BJU Int. 2011 May;107(9):1500-6. doi: 10.1111/j.1464-410X.2010.09555.x. Epub 2010 Aug 24. PMID 20735382
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Background] Phekoo KJ, Schey SA, Richards MA, Bevan DH, Bell S, Gillett D, Moller H; Consultant Haematologists, South Thames Haematology Specialist Committee. A population study to define the incidence and survival of multiple myeloma in a National Health Service Region in UK. Br J Haematol. 2004 Nov;127(3):299-304. doi: 10.1111/j.1365-2141.2004.05207.x. PMID 15491289
- [Background] Sant M, Allemani C, Tereanu C, De Angelis R, Capocaccia R, Visser O, Marcos-Gragera R, Maynadie M, Simonetti A, Lutz JM, Berrino F; HAEMACARE Working Group. Incidence of hematologic malignancies in Europe by morphologic subtype: results of the HAEMACARE project. Blood. 2010 Nov 11;116(19):3724-34. doi: 10.1182/blood-2010-05-282632. Epub 2010 Jul 27. PMID 20664057
- [Background] Smith A, Howell D, Patmore R, Jack A, Roman E. Incidence of haematological malignancy by sub-type: a report from the Haematological Malignancy Research Network. Br J Cancer. 2011 Nov 22;105(11):1684-92. doi: 10.1038/bjc.2011.450. Epub 2011 Nov 1. PMID 22045184
- [Background] Kyle RA, Rajkumar SV. Multiple myeloma. Blood. 2008 Mar 15;111(6):2962-72. doi: 10.1182/blood-2007-10-078022. PMID 18332230
- [Background] Raab MS, Podar K, Breitkreutz I, Richardson PG, Anderson KC. Multiple myeloma. Lancet. 2009 Jul 25;374(9686):324-39. doi: 10.1016/S0140-6736(09)60221-X. Epub 2009 Jun 21. PMID 19541364
- [Background] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015
- [Background] Combination chemotherapy versus melphalan plus prednisone as treatment for multiple myeloma: an overview of 6,633 patients from 27 randomized trials. Myeloma Trialists' Collaborative Group. J Clin Oncol. 1998 Dec;16(12):3832-42. doi: 10.1200/JCO.1998.16.12.3832. PMID 9850028
- [Background] Kumar SK, Lee JH, Lahuerta JJ, Morgan G, Richardson PG, Crowley J, Haessler J, Feather J, Hoering A, Moreau P, LeLeu X, Hulin C, Klein SK, Sonneveld P, Siegel D, Blade J, Goldschmidt H, Jagannath S, Miguel JS, Orlowski R, Palumbo A, Sezer O, Rajkumar SV, Durie BG; International Myeloma Working Group. Risk of progression and survival in multiple myeloma relapsing after therapy with IMiDs and bortezomib: a multicenter international myeloma working group study. Leukemia. 2012 Jan;26(1):149-57. doi: 10.1038/leu.2011.196. Epub 2011 Jul 29. PMID 21799510
- [Background] Liu J, Hamrouni A, Wolowiec D, Coiteux V, Kuliczkowski K, Hetuin D, Saudemont A, Quesnel B. Plasma cells from multiple myeloma patients express B7-H1 (PD-L1) and increase expression after stimulation with IFN-gamma and TLR ligands via a MyD88-, TRAF6-, and MEK-dependent pathway. Blood. 2007 Jul 1;110(1):296-304. doi: 10.1182/blood-2006-10-051482. Epub 2007 Mar 15. PMID 17363736
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Hallett WH, Jing W, Drobyski WR, Johnson BD. Immunosuppressive effects of multiple myeloma are overcome by PD-L1 blockade. Biol Blood Marrow Transplant. 2011 Aug;17(8):1133-45. doi: 10.1016/j.bbmt.2011.03.011. Epub 2011 Apr 12. PMID 21536144
- [Background] Berger R, Rotem-Yehudar R, Slama G, Landes S, Kneller A, Leiba M, Koren-Michowitz M, Shimoni A, Nagler A. Phase I safety and pharmacokinetic study of CT-011, a humanized antibody interacting with PD-1, in patients with advanced hematologic malignancies. Clin Cancer Res. 2008 May 15;14(10):3044-51. doi: 10.1158/1078-0432.CCR-07-4079. PMID 18483370
- [Background] Cavo M, Tacchetti P, Patriarca F, Petrucci MT, Pantani L, Galli M, Di Raimondo F, Crippa C, Zamagni E, Palumbo A, Offidani M, Corradini P, Narni F, Spadano A, Pescosta N, Deliliers GL, Ledda A, Cellini C, Caravita T, Tosi P, Baccarani M; GIMEMA Italian Myeloma Network. Bortezomib with thalidomide plus dexamethasone compared with thalidomide plus dexamethasone as induction therapy before, and consolidation therapy after, double autologous stem-cell transplantation in newly diagnosed multiple myeloma: a randomised phase 3 study. Lancet. 2010 Dec 18;376(9758):2075-85. doi: 10.1016/S0140-6736(10)61424-9. Epub 2010 Dec 9. PMID 21146205
- [Background] Boyd KD, Ross FM, Tapper WJ, Chiecchio L, Dagrada G, Konn ZJ, Gonzalez D, Walker BA, Hockley SL, Wardell CP, Gregory WM, Child JA, Jackson GH, Davies FE, Morgan GJ; NCRI Haematology Oncology Studies Group. The clinical impact and molecular biology of del(17p) in multiple myeloma treated with conventional or thalidomide-based therapy. Genes Chromosomes Cancer. 2011 Oct;50(10):765-74. doi: 10.1002/gcc.20899. PMID 21961181
- [Background] Munshi NC, Anderson KC, Bergsagel PL, Shaughnessy J, Palumbo A, Durie B, Fonseca R, Stewart AK, Harousseau JL, Dimopoulos M, Jagannath S, Hajek R, Sezer O, Kyle R, Sonneveld P, Cavo M, Rajkumar SV, San Miguel J, Crowley J, Avet-Loiseau H; International Myeloma Workshop Consensus Panel 2. Consensus recommendations for risk stratification in multiple myeloma: report of the International Myeloma Workshop Consensus Panel 2. Blood. 2011 May 5;117(18):4696-700. doi: 10.1182/blood-2010-10-300970. Epub 2011 Feb 3. PMID 21292777
- [Background] Palumbo A, Avet-Loiseau H, Oliva S, Lokhorst HM, Goldschmidt H, Rosinol L, Richardson P, Caltagirone S, Lahuerta JJ, Facon T, Bringhen S, Gay F, Attal M, Passera R, Spencer A, Offidani M, Kumar S, Musto P, Lonial S, Petrucci MT, Orlowski RZ, Zamagni E, Morgan G, Dimopoulos MA, Durie BG, Anderson KC, Sonneveld P, San Miguel J, Cavo M, Rajkumar SV, Moreau P. Revised International Staging System for Multiple Myeloma: A Report From International Myeloma Working Group. J Clin Oncol. 2015 Sep 10;33(26):2863-9. doi: 10.1200/JCO.2015.61.2267. Epub 2015 Aug 3. PMID 26240224
- [Background] Neben K, Lokhorst HM, Jauch A, Bertsch U, Hielscher T, van der Holt B, Salwender H, Blau IW, Weisel K, Pfreundschuh M, Scheid C, Duhrsen U, Lindemann W, Schmidt-Wolf IG, Peter N, Teschendorf C, Martin H, Haenel M, Derigs HG, Raab MS, Ho AD, van de Velde H, Hose D, Sonneveld P, Goldschmidt H. Administration of bortezomib before and after autologous stem cell transplantation improves outcome in multiple myeloma patients with deletion 17p. Blood. 2012 Jan 26;119(4):940-8. doi: 10.1182/blood-2011-09-379164. Epub 2011 Dec 8. PMID 22160383
- [Background] Shaughnessy JD Jr, Zhan F, Burington BE, Huang Y, Colla S, Hanamura I, Stewart JP, Kordsmeier B, Randolph C, Williams DR, Xiao Y, Xu H, Epstein J, Anaissie E, Krishna SG, Cottler-Fox M, Hollmig K, Mohiuddin A, Pineda-Roman M, Tricot G, van Rhee F, Sawyer J, Alsayed Y, Walker R, Zangari M, Crowley J, Barlogie B. A validated gene expression model of high-risk multiple myeloma is defined by deregulated expression of genes mapping to chromosome 1. Blood. 2007 Mar 15;109(6):2276-84. doi: 10.1182/blood-2006-07-038430. Epub 2006 Nov 14. PMID 17105813
- [Background] Boyd KD, Ross FM, Chiecchio L, Dagrada GP, Konn ZJ, Tapper WJ, Walker BA, Wardell CP, Gregory WM, Szubert AJ, Bell SE, Child JA, Jackson GH, Davies FE, Morgan GJ; NCRI Haematology Oncology Studies Group. A novel prognostic model in myeloma based on co-segregating adverse FISH lesions and the ISS: analysis of patients treated in the MRC Myeloma IX trial. Leukemia. 2012 Feb;26(2):349-55. doi: 10.1038/leu.2011.204. Epub 2011 Aug 12. PMID 21836613
- [Background] Landgren O, Waxman AJ. Multiple myeloma precursor disease. JAMA. 2010 Dec 1;304(21):2397-404. doi: 10.1001/jama.2010.1713. PMID 21119086
- [Background] Corral LG, Haslett PA, Muller GW, Chen R, Wong LM, Ocampo CJ, Patterson RT, Stirling DI, Kaplan G. Differential cytokine modulation and T cell activation by two distinct classes of thalidomide analogues that are potent inhibitors of TNF-alpha. J Immunol. 1999 Jul 1;163(1):380-6. PMID 10384139
- [Background] Richardson PG, Blood E, Mitsiades CS, Jagannath S, Zeldenrust SR, Alsina M, Schlossman RL, Rajkumar SV, Desikan KR, Hideshima T, Munshi NC, Kelly-Colson K, Doss D, McKenney ML, Gorelik S, Warren D, Freeman A, Rich R, Wu A, Olesnyckyj M, Wride K, Dalton WS, Zeldis J, Knight R, Weller E, Anderson KC. A randomized phase 2 study of lenalidomide therapy for patients with relapsed or relapsed and refractory multiple myeloma. Blood. 2006 Nov 15;108(10):3458-64. doi: 10.1182/blood-2006-04-015909. Epub 2006 Jul 13. PMID 16840727
- [Background] Richardson PG, Mitsiades C, Hideshima T, Anderson KC. Lenalidomide in multiple myeloma. Expert Rev Anticancer Ther. 2006 Aug;6(8):1165-73. doi: 10.1586/14737140.6.8.1165. PMID 16925483
- [Background] Weber DM, Chen C, Niesvizky R, Wang M, Belch A, Stadtmauer EA, Siegel D, Borrello I, Rajkumar SV, Chanan-Khan AA, Lonial S, Yu Z, Patin J, Olesnyckyj M, Zeldis JB, Knight RD; Multiple Myeloma (009) Study Investigators. Lenalidomide plus dexamethasone for relapsed multiple myeloma in North America. N Engl J Med. 2007 Nov 22;357(21):2133-42. doi: 10.1056/NEJMoa070596. PMID 18032763
- [Background] Dimopoulos M, Spencer A, Attal M, Prince HM, Harousseau JL, Dmoszynska A, San Miguel J, Hellmann A, Facon T, Foa R, Corso A, Masliak Z, Olesnyckyj M, Yu Z, Patin J, Zeldis JB, Knight RD; Multiple Myeloma (010) Study Investigators. Lenalidomide plus dexamethasone for relapsed or refractory multiple myeloma. N Engl J Med. 2007 Nov 22;357(21):2123-32. doi: 10.1056/NEJMoa070594. PMID 18032762
- [Background] Richardson PG, Schlossman RL, Weller E, Hideshima T, Mitsiades C, Davies F, LeBlanc R, Catley LP, Doss D, Kelly K, McKenney M, Mechlowicz J, Freeman A, Deocampo R, Rich R, Ryoo JJ, Chauhan D, Balinski K, Zeldis J, Anderson KC. Immunomodulatory drug CC-5013 overcomes drug resistance and is well tolerated in patients with relapsed multiple myeloma. Blood. 2002 Nov 1;100(9):3063-7. doi: 10.1182/blood-2002-03-0996. PMID 12384400
- [Background] Chen C, R.D., Siegel D, et al., Expanded access program (EAP) for lenalidomide plus dexamethasoen in over 1400 subjects with relapsed or refractory multiple myeloma. Blood (ASH Annual Meeting Abstracts), 2006. 108(Abstract 3556).
- [Background] Rajkumar SV, Jacobus S, Callander NS, Fonseca R, Vesole DH, Williams ME, Abonour R, Siegel DS, Katz M, Greipp PR; Eastern Cooperative Oncology Group. Lenalidomide plus high-dose dexamethasone versus lenalidomide plus low-dose dexamethasone as initial therapy for newly diagnosed multiple myeloma: an open-label randomised controlled trial. Lancet Oncol. 2010 Jan;11(1):29-37. doi: 10.1016/S1470-2045(09)70284-0. Epub 2009 Oct 21. PMID 19853510
- [Background] Benboubker L, Dimopoulos MA, Dispenzieri A, Catalano J, Belch AR, Cavo M, Pinto A, Weisel K, Ludwig H, Bahlis N, Banos A, Tiab M, Delforge M, Cavenagh J, Geraldes C, Lee JJ, Chen C, Oriol A, de la Rubia J, Qiu L, White DJ, Binder D, Anderson K, Fermand JP, Moreau P, Attal M, Knight R, Chen G, Van Oostendorp J, Jacques C, Ervin-Haynes A, Avet-Loiseau H, Hulin C, Facon T; FIRST Trial Team. Lenalidomide and dexamethasone in transplant-ineligible patients with myeloma. N Engl J Med. 2014 Sep 4;371(10):906-17. doi: 10.1056/NEJMoa1402551. PMID 25184863
- [Background] Durie BG, Harousseau JL, Miguel JS, Blade J, Barlogie B, Anderson K, Gertz M, Dimopoulos M, Westin J, Sonneveld P, Ludwig H, Gahrton G, Beksac M, Crowley J, Belch A, Boccadaro M, Cavo M, Turesson I, Joshua D, Vesole D, Kyle R, Alexanian R, Tricot G, Attal M, Merlini G, Powles R, Richardson P, Shimizu K, Tosi P, Morgan G, Rajkumar SV; International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006 Sep;20(9):1467-73. doi: 10.1038/sj.leu.2404284. Epub 2006 Jul 20. PMID 16855634
- [Background] Palumbo A, Dimopoulos M, San Miguel J, Harousseau JL, Attal M, Hussein M, Knop S, Ludwig H, von Lilienfeld-Toal M, Sonneveld P. Lenalidomide in combination with dexamethasone for the treatment of relapsed or refractory multiple myeloma. Blood Rev. 2009 Mar;23(2):87-93. doi: 10.1016/j.blre.2008.07.003. Epub 2008 Sep 6. PMID 18774632

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab + Lenalidomide: This is an open label study.
  * Pembrolizumab 200 mg IV every 3 weeks and lenalidomide 25 mg po daily x 14 days and dexamethasone 40 mg po once weekly for a 21-day cycle x 2 cycles.
  * This is followed by pembrolizumab 200 mg every 3 weeks and lenalidomide 25 mg po daily x 14 days for a 21-day cycle x 2 cycles for a total of 4 cycles.
  Pembrolizumab: Pembrolizumab 200 mg IV every 3 weeks x 2 cycles. This is followed by followed by pembrolizumab 200 mg IV every 3 weeks for 2 additional cycles.
  Lenalidomide: Lenalidomide 25 mg po daily x 14 days once weekly for a 21-day cycle x 2 cycles. This is followed by lenalidomide 25 mg po daily x 14 days for a 21-day cycle x 2 cycles for 2 additional cycles.
  Dexamethasone: Dexamethasone 40 mg po once weekly for a 21-day cycle x 2 cycles only.
Period: Overall Study
Arm/Group | Pembrolizumab + Lenalidomide
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab + Lenalidomide
Number analyzed (Participants) | 12
Age, Customized [Mean (Full Range); unit: years]
  Age | 67.2 [63.9 to 70.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10
  Non-White | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS will be assessed from the date of ASCT, with day 0 defined as date of stem cell infusion (if tandem transplant the 2nd of 2 transplants will be used) until the date of progression, defined as the date at which the patient starts the next line of therapy or the date of death.
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: months
Arm/Group | Pembrolizumab + Lenalidomide
Number analyzed (Participants) | 11
months | 27.6 [10 to 30.1]

2. Secondary Outcome: Number of Participants Serious Adverse Events
Description: Safety will be assessed by quantifying the toxicities and grades experienced by subjects who have received pembrolizumab (MK-3475), lenalidomide and dexamethasone, including serious adverse events (SAEs). Result reflects count of participants who experienced an SAE.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenalidomide
Number analyzed (Participants) | 12
Participants | 1

3. Secondary Outcome: Evaluation of Stringent Complete Response, Complete Response, and Very Good Partial Response Rate (sCR + CR + VGPR Rate).
Description: Assessed by the investigator per International Myeloma Working Group criteria(IMWG) uniform response criteria. Result reflects number of participants whose best overall response qualified as sCR, CR, or VGPR in 2 year follow up period.
Time Frame: Every 3 weeks (day 1 of every 21-day treatment cycle +/- 7 days) through 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenalidomide
Number analyzed (Participants) | 11
Participants | 11

4. Secondary Outcome: Number of Participants Who Progressed at 12 Months
Description: Assessed at 12 months; Subjects without documented PD or death will be censored at the last disease assessment date. Those who died without documented PD will be censored at the time of death. Result reflects count of participants who had progressed at 12 months.
Time Frame: Time from Day 0 (transplant) and date of enrollment to study completion (through 12 weeks) by investigator assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Lenalidomide
Number analyzed (Participants) | 11
Participants | 10

5. Secondary Outcome: Duration of Response (DOR)
Description: Assessed by the investigator per International Myeloma Working Group criteria(IMWG) uniform response criteria. Result reflects count of participants who did not have progressive disease at 2 years.
Time Frame: Interval between date of first response and date of study completion (through 12 weeks)
Population: The FDA required enrollment to stop and patients to be removed from treatment due to updated risks of the investigational product. Following removal of the study data was not collected and patients were not analyzed due to this early termination of study intervention.
Arm/Group | Pembrolizumab + Lenalidomide
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Comparison in Bone Marrow Aspirates of the Extent of Pre-pembrolizumab (MK-3475), Lenalidomide and Dexamethasone PD-L1 Expression and Change From Baseline PD-L1 Expression in Responders Versus Non-responders
Description: Comparison of change from baseline in bone marrow aspirate/biopsy PD-L1 expression between responders with longer duration of response and non-responders or responders with a short duration of response will be performed using mixed regression analysis. Longitudinal analysis of bone marrow aspirate/biopsy PD-L1 expression over time will be examined using mixed model repeated measure design with levels observed serially over time and response type (long responders vs short responders/non-response) as a fixed variable.
Time Frame: Bone marrow aspirate specimens will be obtained at screening and at week 15 (completion of cycle 4).
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Assessment of Immune Phenotype in Bone Marrow Aspirates and Peripheral Blood Samples and Plasma Cytokines.
Description: Assays for these studies include flow cytometry, TCR Immunoseq for Vbeta CDR3 highest frequency specificities, real-time PCR analysis and multiplex cytokine ELISA. These data will be aggregated before and after treatment in responders versus non-responders.
Time Frame: Obtained monthly through week 12 (cycle 4 day 1).
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Assessment of T Cell Repertoire in Bone Marrow Aspirates and Peripheral Blood Samples.
Description: Assays for these studies include flow cytometry, TCR Immunoseq for Vbeta CDR3 highest frequency specificities, and real-time PCR analysis. T cells (CD8+) data will be aggregated before and after treatment in responders versus non-responders.
Time Frame: Obtained monthly through week 12 (cycle 4 day 1).
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Assessment of Plasma Cytokines
Description: Multiplex cytokine ELISA studies will assess inflammatory cytokine (TNF-alpha, IL-2, IL-4, IL-6, IL-10) data and will be aggregated before and after treatment in responders versus non-responders.
Time Frame: Obtained monthly through week 12 (cycle 4 day 1).
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Identification and Assessment of Specific Intestinal Microbial Strains (Via Stool Specimens) Associated With Improved Outcome in Autologous Stem Cell Transplantation Patients Treated With PEM+LEN+DEX Compared to PEM+LEN.
Description: A 16S ribosomal RNA (rRNA) miSeq Illumina platform will be used for overall microbial composition and quantitative real-time PCR analysis will validate the specific microbial strains identified by miSeq.
Time Frame: Stool specimens at screening or cycle 1, day 1, cycle 2 day 1, cycle 3 day 1, cycle 4 day 1, at completion of cycle 4, and at 90 days post treatment or start of new anti cancer therapy. Stool samples will also be collected at confirmation of response.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Study Enrollment to Study Completion, up to 3 years
Arm/Group | Pembrolizumab + Lenalidomide
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenalidomide (N=12)
H. Influenza Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Lenalidomide (N=12)
Neutropenia (Blood and lymphatic system disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Fatigue (Psychiatric disorders) | 1
Increased ALT (Blood and lymphatic system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT02906332/Prot_SAP_000.pdf